CLINICAL TRIAL: NCT00583284
Title: Utility of Delayed-Enhancement Multi-Detector Computed Tomography Imaging in Identifying Arrhymogenic Substrate in Patients Undergoing Catheter Ablation for Ventricular Tachycardia
Brief Title: The Use of CT to Identify Damaged Heart Muscle in Patients Undergoing Ventricular Tachycardia Ablation.
Status: Terminated | Type: Observational
Why Stopped: key study staff left foundation
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 06-647
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Ventricular Tachycardia
Keywords: delayed enhancement computed tomography; ventricular tachycardia ablation; ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with ventricular tachycardia (VT) undergo catheter ablation. During the ablation procedure, the heart is mapped to determine areas of heart muscle damage. The heart scarring areas are often the source of the VT. Delayed enhancement CT has recently been used to determine areas of scarring . This study is to determine if the areas of damaged heart muscle mapped with the delayed enhancement CT correlate with the same areas that are determined during the catheter ablation.

DETAILED DESCRIPTION:
Catheter ablation of ventricular tachycardia (VT) is performed in patients who have recurrent VT despite the use of other therapies. Electroanatomic mapping of the left ventricular myocardium is performed as part of these procedures to define the arrhythmogenic substrate for subsequent ablation. We hypothesize that delayed enhancement multi-detector computed tomography (MDCT) will identify areas of myocardial scarring or fibrosis that correlate with findings of voltage mapping in patients with a prior myocardial infarction who are undergoing VT ablation. We will perform a pilot study involving 10 patients with coronary artery disease scheduled for VT ablation to determine the ability of delayed enhancement MDCT to identify arrhythmogenic substrates in these patients, when compared with electroanatomic mapping. All patients will undergo a standard of care 64-slice MDCT study, followed 5 minutes later by the research delayed enhancement acquisition. We will evaluate the relationship between hyperenhanced myocardium, as detected by delayed enhancement MDCT, and abnormal myocardium detected on voltage mapping, defined as areas of myocardium with < 0.5 mV signal amplitude. Studies will be performed on the new Siemens 64-slice dual source CT scanner, which reduces radiation exposure from the scan by 33-50%. This study will generate preliminary data which will be used for subsequent NIH/AHA grant applications or industry sponsored trials.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Prior myocardial infarction
* Scheduled for CT scan < 1 week prior to VT ablation for ventricular arrythmia

Exclusion Criteria:

* Serum creatinine > 1.8 mg/dL
* Contrast dye allergy
* Atrial fibrillation
* Unable to lie flat for the duration of image acquistion (15-20 minutes)
* Clinical instability at time of CT study acquisition
* Women of childbearing potential
* Personal or social problems that might prevent compliance with the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming to Cleveland Clinic for catheter ablation for ventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Areas of hyperenhanced myocardium, as determined by delayed enhancement CT, correlate with the findings on voltage mapping of the LV in patients with a prior myocardial infarction who are undergoing VT ablation. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Srikanth Sola, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226